CLINICAL TRIAL: NCT05501899
Title: Use of Levocarnitine to Reduce Asparaginase Hepatotoxicity in Patients With Acute Lymphoblastic Leukemia
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Children's Hospital of Orange County (Other)
Collaborators: University of California, Irvine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2110145
Record Dates: First submitted 2022-08-12; First posted 2022-08-16 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Acute Lymphoblastic Leukemia; Hepatotoxicity
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Carnitine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm (single arm) (Experimental)
  Interventions: Drug: Levocarnitine

INTERVENTIONS:
Drug: Levocarnitine — Adults, or patients ≥ 50 kg: 990 mg PO (by mouth) bis in die (BID, twice a day) Children, or patients < 50 kg: 50 mg/kg/day PO divided BID (maximum daily dose of 2,000 mg)
  Other Names: Carnitor®

SUMMARY:
Acute lymphoblastic leukemia (ALL) is the most common cancer seen in pediatric oncology. The necessary chemotherapy for pediatric and adolescent and young adult (AYA) patients with ALL includes steroids, anthracyclines, asparaginase, and vincristine. One of the most hepatotoxic chemotherapy agents is asparaginase, with treatment-associated hepatotoxicity (TAH) observed in up to 60% of patients. The frequency of TAH is increased in overweight or obese patients of Latino heritage. Carnitine is a naturally-derived compound that is produced in the liver and kidneys; it is found in certain foods, such as meat, poultry, fish, and some dairy products. Endogenous carnitine transports long-chain fatty acids into the mitochondria, where they are oxidized to produce energy, and acts as scavengers of oxygen free radicals. Thus, carnitine can reduce oxidative stress and modulate inflammatory response. Levocarnitine is a supplement form of carnitine used typically in the care and management of patients with carnitine deficiency. Pediatric and AYAs with ALL will be given oral levocarnitine as a supplement during their initial phases of treatment, when the most hepatotoxic agents are administered, to determine if the incidence of liver toxicity can be reduced or eliminated.

DETAILED DESCRIPTION:
Primary Aims

1. Prospectively evaluate whether the prophylactic use of levocarnitine during Induction and Consolidation (phases with asparaginase therapy) in ALL patients receiving treatment according to a Children's Oncology Group (COG) treatment protocol reduces hepatotoxicity.
2. Demonstrate an association between ethnicity and liver function test abnormalities in children and AYAs with ALL. Specifically, that Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 grade ≥ 3 elevated liver function tests is more prevalent in self-identified Latinos as compared to other ethnicities in a retrospective control group.

Secondary Aims

1. Determine whether obesity or overweight status, as measured by body mass index, at diagnosis increases the risk of hepatic dysfunction.
2. Quantify the disease response, based on the end of Induction minimal residual disease (MRD) in the bone marrow of patients receiving levocarnitine, compared to historical controls to determine that levocarnitine does not have a negative impact on MRD.
3. Assess incidence of nonalcoholic fatty liver disease (NAFLD), via non-invasive ultrasound elastography, in pediatric and AYA patients newly diagnosed with ALL.
4. Assess incidence of other known toxicities of asparaginase treatment, including hyper/hypoglycemia, hypertriglyceridemia, pancreatitis, and thrombosis that are CTCAE version 5.0 grade ≥ 3 with onset ≤ 30 days (or next dose if sooner) of asparaginase.

Study Design:

The proposal is a non-randomized case-control pilot study that will use retrospective case-control data as comparison (i.e., control group).

Participants:

A sample of 20 pediatric and AYA patients, ages 5 to < 30 years, newly diagnosed with ALL will be enrolled to study. Participants who withdraw or who are withdrawn from study, who have taken less than 50% of planned levocarnitine supplementation, and who did not have a post-levocarnitine supplementation laboratory testing will be replaced. An additional 20 retrospective cases -- matched by age at diagnosis, biological sex, and risk classification at initial diagnosis -- will be included to provide control data.

Study Intervention:

Levocarnitine will be administered by mouth twice daily during Induction and Consolidation phases of treatment for patients with ALL who are treated as per a COG treatment plan (either on study or treated according to the protocol). The duration of intervention is expected to be approximately three months.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 5 to < 30 years
* Newly diagnosed with ALL designated as NCI high-risk (HR) ALL
* Treatment for ALL to be according to a Children's Oncology Group (COG) treatment protocol (on study or according to study)
* Ability to take oral medications and willing to adhere to the levocarnitine regimen

Exclusion Criteria:

* Known allergic reaction to levocarnitine or its components
* Presence of severely compromised renal function or end-stage renal disease
* Pregnancy or lactation
* Warfarin therapy
* History of seizures prior to ALL diagnosis
* Known inborn error of metabolism

Ages: 5 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-03-03 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome #1 | 1.5 years
  Calculate proportion of patients who experience hepatotoxicity, as measured by the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 grade ≥ 3 elevated alanine aminotransferase (ALT), aspartate aminotransferase (AST), and total and direct bilirubin.
Primary Outcome #2 | 1.5 years
  Calculate prevalence of hepatotoxicity in patients who self-identify as Latino or non-Latino, using laboratory assessments and self-reported measures of ethnicity and/or race.

SECONDARY OUTCOMES:
Secondary Outcome #1 | 1.5 years
  Calculate body mass index (BMI), from recorded height and weight obtained at time of initial diagnosis and determine if there is increased risk of hepatotoxicity in patients who are overweight or obese at diagnosis as determined by Centers for Disease Control and Prevention (CDC) clinical growth charts for study participants 5 to < 20 years of age and by a BMI of ≥ 25.0 for study participants 20 to < 30 years of age.
Secondary Outcome #2 | 1.5 years
  Quantify disease response, using end of Induction minimal residual disease (MRD) results, where an MRD value < 0.01 is considered "negative."
Secondary Outcome #3 | 1.5 years
  Calculate incidence of nonalcoholic fatty liver disease (NAFLD), using ultrasound elastography, in pediatric and AYA patients newly diagnosed with ALL.
Secondary Outcome #4 | 1.5 years
  Calculate proportion of patients who experience other known toxicities of asparaginase treatment, as measured by CTCAE version 5.0 grade ≥ 3 hyper/hypoglycemia, hypertriglyceridemia, pancreatitis, and thrombosis.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Chao Family Comprehensive Cancer Center, University of California, Irvine, Orange, California
  - Children's Hospital of Orange County, Orange, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hunger SP, Lu X, Devidas M, Camitta BM, Gaynon PS, Winick NJ, Reaman GH, Carroll WL. Improved survival for children and adolescents with acute lymphoblastic leukemia between 1990 and 2005: a report from the children's oncology group. J Clin Oncol. 2012 May 10;30(14):1663-9. doi: 10.1200/JCO.2011.37.8018. Epub 2012 Mar 12. PMID 22412151
- [Background] Kadan-Lottick NS, Ness KK, Bhatia S, Gurney JG. Survival variability by race and ethnicity in childhood acute lymphoblastic leukemia. JAMA. 2003 Oct 15;290(15):2008-14. doi: 10.1001/jama.290.15.2008. PMID 14559954
- [Background] DeAngelo DJ, Stevenson KE, Dahlberg SE, Silverman LB, Couban S, Supko JG, Amrein PC, Ballen KK, Seftel MD, Turner AR, Leber B, Howson-Jan K, Kelly K, Cohen S, Matthews JH, Savoie L, Wadleigh M, Sirulnik LA, Galinsky I, Neuberg DS, Sallan SE, Stone RM. Long-term outcome of a pediatric-inspired regimen used for adults aged 18-50 years with newly diagnosed acute lymphoblastic leukemia. Leukemia. 2015 Mar;29(3):526-34. doi: 10.1038/leu.2014.229. Epub 2014 Jul 31. PMID 25079173
- [Background] Stock W, Luger SM, Advani AS, Yin J, Harvey RC, Mullighan CG, Willman CL, Fulton N, Laumann KM, Malnassy G, Paietta E, Parker E, Geyer S, Mrozek K, Bloomfield CD, Sanford B, Marcucci G, Liedtke M, Claxton DF, Foster MC, Bogart JA, Grecula JC, Appelbaum FR, Erba H, Litzow MR, Tallman MS, Stone RM, Larson RA. A pediatric regimen for older adolescents and young adults with acute lymphoblastic leukemia: results of CALGB 10403. Blood. 2019 Apr 4;133(14):1548-1559. doi: 10.1182/blood-2018-10-881961. Epub 2019 Jan 18. PMID 30658992
- [Background] Aldoss I, Douer D, Behrendt CE, Chaudhary P, Mohrbacher A, Vrona J, Pullarkat V. Toxicity profile of repeated doses of PEG-asparaginase incorporated into a pediatric-type regimen for adult acute lymphoblastic leukemia. Eur J Haematol. 2016 Apr;96(4):375-80. doi: 10.1111/ejh.12600. Epub 2015 Jun 25. PMID 26095294
- [Background] Raetz EA, Salzer WL. Tolerability and efficacy of L-asparaginase therapy in pediatric patients with acute lymphoblastic leukemia. J Pediatr Hematol Oncol. 2010 Oct;32(7):554-63. doi: 10.1097/MPH.0b013e3181e6f003. PMID 20724951
- [Background] Ogden CL, Carroll MD, Kit BK, Flegal KM. Prevalence of childhood and adult obesity in the United States, 2011-2012. JAMA. 2014 Feb 26;311(8):806-14. doi: 10.1001/jama.2014.732. PMID 24570244
- [Background] van der Sluis IM, Vrooman LM, Pieters R, Baruchel A, Escherich G, Goulden N, Mondelaers V, Sanchez de Toledo J, Rizzari C, Silverman LB, Whitlock JA. Consensus expert recommendations for identification and management of asparaginase hypersensitivity and silent inactivation. Haematologica. 2016 Mar;101(3):279-85. doi: 10.3324/haematol.2015.137380. PMID 26928249
- [Background] Romano M, Vacante M, Cristaldi E, Colonna V, Gargante MP, Cammalleri L, Malaguarnera M. L-carnitine treatment reduces steatosis in patients with chronic hepatitis C treated with alpha-interferon and ribavirin. Dig Dis Sci. 2008 Apr;53(4):1114-21. doi: 10.1007/s10620-007-9983-1. Epub 2007 Oct 16. PMID 17939042
- [Background] Schulte RR, Madiwale MV, Flower A, Hochberg J, Burke MJ, McNeer JL, DuVall A, Bleyer A. Levocarnitine for asparaginase-induced hepatic injury: a multi-institutional case series and review of the literature. Leuk Lymphoma. 2018 Oct;59(10):2360-2368. doi: 10.1080/10428194.2018.1435873. Epub 2018 Feb 12. PMID 29431566
- [Background] Aldoss I, Douer D. How I treat the toxicities of pegasparaginase in adults with acute lymphoblastic leukemia. Blood. 2020 Mar 26;135(13):987-995. doi: 10.1182/blood.2019002477. PMID 31977001
- [Background] Schulte R, Hinson A, Huynh V, Breese EH, Pierro J, Rotz S, Mixon BA, McNeer JL, Burke MJ, Orgel E. Levocarnitine for pegaspargase-induced hepatotoxicity in older children and young adults with acute lymphoblastic leukemia. Cancer Med. 2021 Nov;10(21):7551-7560. doi: 10.1002/cam4.4281. Epub 2021 Sep 16. PMID 34528411
- See also: SEER Cancer Statistics Review, 1975-2011 — https://seer.cancer.gov/archive/csr/1975_2011/